CLINICAL TRIAL: NCT03824665
Title: Nalbuphine, Fentanyl and no Additive to Local Anaesthetic Mixture for Peribulbar Block During Posterior Segment Surgery in Adult Patients a Prospective Randomized Clinical Trial
Brief Title: Nalbuphine, Fentanyl and no Additive to Local Anaesthetic Mixture
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Abdalla, Professor of Anesthesia &I.C.U and Pain Clinic, Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Nalbuphine Versus Fentanyl
Record Dates: First submitted 2019-01-19; First posted 2019-01-31 (Actual); Last update posted 2019-05-21 (Actual); Status verified 2019-05

CONDITIONS: Nalbuphine,Fentanyl and Local Anesthetic Mixture
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Evaluation of the analgesic and hemodynamic outcome of nalbuphine or fentanyl versus a control group for peribulbar block (PBB) during posterior chamber surgery.
Who Masked: Participant, Investigator
Masking Description: Patients were grouped randomly using sealed envelopes prepared by an assistant who was blinded to the grouping and envelops were chosen by patient him/her self or by the nearest relative All patients received 8 ml of LAM which consisted of: 3 ml of mepivacaine 3%,
  1 ml of hyaluronidase containing 150 IU, 2 ml of bupivacaine 0.5%, 1 ml of lidocaine 2%.Patients were categorized into three groups according to the type of additive used with the LAM as follows:
  1. Group C (Control group): included patients assigned to receive 1 ml normal saline.
  2. Group F: 1 ml saline containing 20 μg fentanyl was used instead of normal saline.
  3. Group N:1 ml saline containing 4mg nalbuphine was used instead of normal saline.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Nalbuphine Group (Active Comparator): Nalbuphine Group (Nalbuphine) 8 ml of LAM which consisted of: 6 ml of bupivacaine 0.5%, 1 ml of hyaluronidase containing 150 IU, plus 1 ml saline containing 4mg nalbuphine
  Interventions: Drug: Nalbuphine Group
- Fentanyl Group (Active Comparator): Fentanyl Group 8 ml of LAM which consisted of: 6 ml of bupivacaine 0.5%, 1 ml of hyaluronidase containing 150 IU, plus 1 ml saline containing 20 μg fentanyl
  Interventions: Drug: Fentanyl Group
- Control group (Active Comparator): Control group 8 ml of LAM which consisted of: 6 ml of bupivacaine 0.5%, 1 ml of hyaluronidase containing 150 IU, plus 1 ml normal saline
  Interventions: Drug: Control Group

INTERVENTIONS:
Drug: Nalbuphine Group — All patients received 8 ml of LAM which consisted of: 6 ml of ml of bupivacaine 0.5%, 1 ml of hyaluronidase containing 150 IU, 1 ml of additive
  Patients were categorized into three groups according to the type of additive used with the LAM as follows:
  Group N:(Nalbuphine group)1 ml saline containing 4mg nalbuphine used instead of normal saline
  Other Names: Group N
  Arms: Nalbuphine Group
Drug: Fentanyl Group — All patients received 8 ml of LAM which consisted of: 6 ml of ml of bupivacaine 0.5%, 1 ml of hyaluronidase containing 150 IU, 1 ml of additive
  Patients were categorized into three groups according to the type of additive used with the LAM as follows:
  Group F: :(Fentanyl group)1 ml saline containing 20 μg fentanyl used instead of normal saline
  Other Names: Group F
  Arms: Fentanyl Group
Drug: Control Group — All patients received 8 ml of LAM which consisted of: 6 ml of ml of bupivacaine 0.5%, 1 ml of hyaluronidase containing 150 IU, 1 ml of additive
  Patients were categorized into three groups according to the type of additive used with the LAM as follows:
  Group C (Control group): included patients assigned to receive 1 ml normal saline.
  Other Names: Group C
  Arms: Control group

SUMMARY:
Nalbuphine has been used as an adjuvant to bupivacaine in intrathecal,epidural, caudal anesthesia and peripheral nerve blocks showing an increase in the efficacy and the duration of postoperative analgesia. The aim of this study is evaluation of the effect of 4 mg Nalbuphine when used as an adjuvant to a local anesthetic mixture in peribulbar block undergoing posterior chamber surgery in adult patients and comparing it with adding Fentanyl 20 μg to LAM and LAM alone

DETAILED DESCRIPTION:
120 patients (40 in each group) scheduled for elective posterior chamber surgery using peribulbar block. Patients of Group N received 6 ml of 0.5% bupivacaine 1 ml hyaluronidase (75 IU), and 4mg of Nalbuphine in 1 ml of saline (total 8 ml) and patients of Group F received 6 ml of 0.5% bupivacaine 6 ml of 0.5% bupivacaine 1 ml hyaluronidase (75 IU), and 20 μg fentanyl in 1 ml saline (total 8 ml) and Group C received 6 ml of 0.5% bupivacaine,1 ml hyaluronidase (75 IU) and1 ml saline (total 8 ml).

Study outcomes included evaluation and scoring (onset and duration) of eyelid and globe akinesia, total 15-min akinesia score and duration of block.

Intraoperative hemodynamic measures were measured every 15 minutes during the whole procedure and every 30 minutes during the first two postoperative (PO) hours.. PO analgesia was hourly-assessed using Visual Analogue Score (VAS) and analgesia was provided at VAS of >5.

Anesthetic procedure After securing intravenous access, non-invasive monitoring for blood pressure (SBP, DBP, MAP), E.C.G, and pulse oximetry (SpO2) were applied. tetracaine eye drops 0.5% applied to all patients as topical anesthesia. All patients were sedated using midazolam (0.05 mg/kg) as a preanesthetic medication I.V prior to receive LAM injection with nasal oxygen mask. Two ml of lidocaine 2% were diluted with 8 ml saline 3ml of LAM assigned for each group was injected in the medial canthus (the tunnel between the caruncle and the medial canthal angle) using needle 3-cm length and 27G inserted at angle of 45° between the caruncle and medial canthal angle till the tip of the needle touch the ethmoid bone then the direction of the needle was changed to 90° with the hub of the needle at level of the iris. Another 5 ml of LAM was injected at the extreme inferotemporal border of the orbit with the same needle directed downward and medially below the globe. Light orbital compression applied for 1 minute; then eye was evaluated 1, 3, 5 and 10 minutes for appearance of proptosis and chemosis.

All patients receive intraoperative non-invasive monitoring for blood pressure measures (SBP, DBP, MAP),E.C.G, and pulse oximetry (SpO2) prior to local anesthetic injection.

ELIGIBILITY:
Inclusion Criteria:

* patients aged 40-70 years.
* both sex.
* ASA physical status Ι&II.
* Patient with axial globe length below 26

Exclusion Criteria:

* Refusal of the patient to participate in the study.
* Coagulation abnormalities(INR>1.4).
* More than ASA II.
* High myopia with axial length more than 26 mm.
* Mentally retarded patients and failure of proper communication as in deafness .
* Morbidly obese patients(BMI>35)
* Patients with glaucoma (increased IOP>20mmgh)
* Patients with history of hypersensitivity to study drugs

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2019-02-05 (Actual); Primary Completion 2019-05-10 (Actual); Study Completion 2019-05-18 (Actual)

PRIMARY OUTCOMES:
Onset of eyelid and globe akinesia | 24 hours Postoperative
  The onset of eyelid and globe akinesia was assessed till complete recovery

SECONDARY OUTCOMES:
Blood pressure | 24 hours Postoperative
  Blood pressure (mmHg) .Hypotension is defined as a 20% decrease in MAP in relation to baseline measures
Heart rate | 24 hours Postoperative
  Heart rate (beat/minute).Bradycardia were defined as a 20% decrease in HR in relation to baseline measures
Post Operative analgesia | 24 hours Postoperative
  Assessed by using 11-points Visual Analogue Score (VAS) every hour for 6-hrs PO and was scored as 0 if no pain up to 10 which indicates sever pain sensation. PO analgesia was provided as if VAS was >5 in the form of I.M injection of pethidine50 mg

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Abdalla Mohamed, M.D, Principal Investigator — Cairo University
Locations (1):
- Ahmed Abdalla Mohamed, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
Till Press